CLINICAL TRIAL: NCT02391805
Title: A Multiple-Center, Randomized, Partially Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antiviral Effects of 12-Week Treatment With RO6864018 in Virologically Suppressed Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study of Treatment With RO6864018 in Virologically Suppressed Participants With Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP28938
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Placebo, Every Other Day (QOD) (Placebo Comparator): Placebo orally (PO) QOD for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: Placebo; Drug: Tenofovir
- Placebo, Once a Week (QWk) (Placebo Comparator): Placebo PO QWk for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: Placebo; Drug: Tenofovir
- RO6864018, 1200 milligrams (mg) QOD (Experimental): RO6864018 1200 mg PO QOD for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: RO6864018; Drug: Tenofovir
- RO6864018, 1200 mg QWk (Experimental): RO6864018 1200 mg PO QWk for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: RO6864018; Drug: Tenofovir
- RO6864018, 800 mg QOD (Experimental): RO6864018 800 mg PO QOD for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: RO6864018; Drug: Tenofovir
- RO6864018, 800 mg QWk (Experimental): RO6864018 800 mg PO QWk for 12 weeks + noninvestigational entecavir or tenofovir as prescribed by participant's physician
  Interventions: Drug: Entecavir; Drug: RO6864018; Drug: Tenofovir

INTERVENTIONS:
Drug: Entecavir — Entecavir will be administered as per local labeling.
Drug: Placebo — Participants will be administered PO placebo capsules matched to RO6864018, either QOD or QWk for 12 weeks of treatment.
  Arms: Placebo, Every Other Day (QOD); Placebo, Once a Week (QWk)
Drug: RO6864018 — Participants will be administered RO6864018 as 200-mg PO capsules at a dose of 800 mg or 1200 mg, either QOD or QWk for 12 weeks of treatment.
  Arms: RO6864018, 1200 mg QWk; RO6864018, 1200 milligrams (mg) QOD; RO6864018, 800 mg QOD; RO6864018, 800 mg QWk
Drug: Tenofovir — Tenofovir will be administered as per local labeling.

SUMMARY:
This randomized, multicenter, partially double-blind, placebo-controlled study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antiviral effects of treatment with RO6864018 in virologically suppressed participants with chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B infection
* Positive test for HBsAg for more than 6 months prior to randomization
* HBsAg titer greater than or equal to (>/=) 250 international units per milliliter (IU/mL) at Screening
* Treatment with any nucleoside/nucleotide analogue for >/= 1 year with ongoing entecavir and/or tenofovir treatment at randomization and for at least 3 months prior to randomization
* HBV DNA less than (<) 90 IU/mL for at least the preceding 6 months
* HBeAg positive at randomization and for at least 6 months prior to randomization

Exclusion Criteria:

* Pregnant or lactating women
* Documented history of HBV genotype D
* History or other evidence of bleeding from esophageal varices
* History of decompensated liver disease, chronic liver disease other than HBV infection, or any evidence of metabolic liver disease
* Positive test for hepatitis A, hepatitis C, or human immunodeficiency virus (HIV)
* Documented history of hepatitis D infection
* History of or suspicion of hepatocellular carcinoma
* History of immunologically mediated disease
* History of organ transplantation
* History of thyroid disease
* Significant acute infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05-17 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Safety: Percentage of Participants with Adverse Events | Baseline up to approximately 36 weeks

SECONDARY OUTCOMES:
Pharmacodynamics: Peripheral Blood Levels of Interferon (IFN)-Alpha in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IFN-Alpha in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IFN-Gamma-Induced Protein (IP)-10 in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IP-10 in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Quantitative HBV Deoxyribonucleic Acid (DNA) Level in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Weeks 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up; and at any point that breakthrough occurs (up to 36 weeks)
Efficacy: Quantitative HBV DNA Level in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up; and at any point that breakthrough occurs (up to 36 weeks)
Efficacy: Quantitative Hepatitis B Surface Antigen (HBsAg) Level in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Weeks 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Quantitative HBsAg Level in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Loss of HBsAg in QOD Dosing Cohorts | Baseline; on Day 7 of Week 12; then at Week 36 during follow-up
Efficacy: Percentage of Participants with Loss of HBsAg in QWk Dosing Cohorts | Baseline; on Day 7 of Week 12; then at Week 36 during follow-up
Efficacy: Percentage of Participants with Loss of Hepatitis B Envelope Antigen (HBeAg) in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Weeks 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Loss of HBeAg in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with HBsAg Seroconversion in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Week 5; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
  HBsAg Seroconversion = antibody to HBsAg (Anti-HBs) Positive Status and Loss of HBsAg
Efficacy: Percentage of Participants with HBsAg Seroconversion in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 5; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
  HBsAg Seroconversion = anti-HBs Positive Status and Loss of HBsAg
Efficacy: Percentage of Participants with HBeAg Seroconversion in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Week 5; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
  HBeAg Seroconversion = antibody to HBeAg (anti-HBe) Positive Status and Loss of HBeAg
Efficacy: Percentage of Participants with HBeAg Seroconversion in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 5; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
  HBeAg Seroconversion = anti-HBe Positive Status and Loss of HBeAg
Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of RO6864018 Metabolite in QOD Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Days 1, 7 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 3, 5, 7, 12 and Day 6 of Week 12
Pharmacokinetics: Cmax of RO6864018 Metabolite in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacokinetics: Time to Maximum Observed Plasma Concentration (Tmax) of RO6864018 Metabolite in QOD Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Days 1, 7 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 3, 5, 7, 12 and Day 6 of Week 12
Pharmacokinetics: Tmax of RO6864018 Metabolite in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacokinetics: Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUCinf) of RO6864018 Metabolite in QOD Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Days 1, 7 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 3, 5, 7, 12 and Day 6 of Week 12
Pharmacokinetics: AUCinf of RO6864018 Metabolite in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacokinetics: Area Under the Plasma Concentration-Time Curve up to the Last Measurable Concentration (AUClast) of RO6864018 Metabolite in QOD Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Days 1, 7 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 3, 5, 7, 12 and Day 6 of Week 12
Pharmacokinetics: AUClast of RO6864018 Metabolite in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacokinetics: Half-life (t1/2) of RO6864018 Metabolite in QOD Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Days 1, 7 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 3, 5, 7, 12 and Day 6 of Week 12
Pharmacokinetics: T1/2 of RO6864018 Metabolite in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacodynamics: Peripheral Blood Levels of Neopterin in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of Neopterin in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of Tumor Necrosis Factor (TNF)-Alpha in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of TNF-alpha in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of Interleukin (IL)-6 in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IL-6 in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IL-10 in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IL-10 in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IL-12p40 in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Days 1, 3, 7 of Week 1; on Day 1 of Weeks 3, 5, 7; and Day 6 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Peripheral Blood Levels of IL-12p40 in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) and post-dose (6, 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Development of Anti-HBe in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Weeks 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Development of Anti-HBe in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Development of Anti-HBs in QOD Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 7 of Week 1 and Day 1 of Weeks 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Efficacy: Percentage of Participants with Development of Anti-HBs in QWk Dosing Cohorts | Baseline; pre-dose (0 hours) on Day 1 of Weeks 2, 3, 5, 7; on Day 7 of Week 12; then at Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Transcriptional Responses as Measured by messenger ribonucleic acid (mRNA) Levels for QWk Cohorts | QWk: Baseline; pre-dose (0 hours) and post-dose (6 and 24 hours) on Day 1 of Weeks 1, 2, 3, 5, 7, 12, and Day 7 of Week 12; then Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Transcriptional Responses as Measured by messenger ribonucleic acid (mRNA) Levels for QOD Cohorts | Baseline; pre-dose; post-dose (6 and 24 hours) on Days 1, 3, and 7 for Week 1, Day 1 of Weeks 3, 5, 7, Day 6 of Week 12; then Weeks 16, 20, 24, 28, 32, 36 during follow-up
Pharmacodynamics: Percentage of T Cells, B Cells, and NK Cells (TBNK) | For QOD and QWk Cohorts: Baseline; pre-dose (0 hours) on Day 1 of Weeks 1, 2, 5; then Weeks 20, 28, 36 during follow-up
Pharmacodynamics: Percentage of Myeloid Cells | For QOD and QWk Cohorts: Baseline; pre-dose (0 hours) on Day 1 of Weeks 1, 2, 5; then Weeks 20, 28, 36 during follow-up
Pharmacodynamics: Percentage of Plasmacytoid Dendritic Cells | For QOD and QWk Cohorts: Baseline; pre-dose (0 hours) on Day 1 of Weeks 1, 2, 5; then Weeks 20, 28, 36 during follow-up
Pharmacokinetics: Cmax of Entecavir in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12
Pharmacokinetics: AUCinf of Entecavir in QWk Dosing Cohorts | Pre-dose (0 hours) and post-dose (0.25, 1, 2, 4, 6, 8, 12, 24 hours) on Day 1 of Week 1; pre-dose (0 hours) and post-dose (1, 2-4 hours) on Day 1 of Weeks 2, 3, 5, 7, 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital; Special Medical Clinic, N.T.
- Malaysia (3):
  - Hospital Ampang, Ampang
  - Hospital Selayang; Medicine, Batu Caves
  - University Malaya Medical Center, Kuala Lumpur
- New Zealand (2):
  - Auckland Clinical Studies Limited, Grafton
  - Waikato Hospital, Hamilton
- Changi General Hospital, Singapore, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (3):
  - Kaohsiung Medical Uni Chung-Ho Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei